CLINICAL TRIAL: NCT00160745
Title: A Randomised, Double-blind, Placebo-controlled, Mono-centre, Explorative Phase II Trial to Study the Effects of Rosuvastatin on Basal Production and Release of Nitric Oxide From the Renal Vasculature in Patients With Hypercholesterolemia.
Brief Title: Rosuvastatin and Renal Endothelial Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Rosuvastatin-study
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hypercholesterolemia
Keywords: endothelium, NO, renal, statins
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
The endothelium plays an important role in the regulation of vascular tone and regulation of blood flow. Nitric oxide (NO) is the most important known endothelium-derived vasodilating factor. Prospective studies have shown that hypercholesterolemia impairs endothelial function in different vascular beds. Lowering total cholesterol and particularly LDL-cholesterol with statins leads to an improvement in endothelium-dependent vasodilation in the forearm vasculature. There is strong evidence to suggest that the benefit is not merely related to the decrease in cholesterol-levels. A recent study in the forearm vasculature demonstrated that short-term lipid-lowering therapy improves endothelial function and NO availability already after 3 days of lipid lowering therapy. Whether endothelial function in the renal vasculature of hypercholesterolemic patients is similarly influenced has not yet been addressed adequately. In the present study we investigate whether lipid lowering therapy with rosuvastatin alters renal endothelial function, as assessed by systemic infusion of the NO synthase inhibitor L-NMMA, after 3 and 42 days of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged between 18 and 75 years
* fasting LDL C concentrations >=160 and < 250mg/dl
* fasting TG concentrations =< 350mg/dl

Exclusion Criteria:

* History of statin induced myopathy, or serious hypersensitivity reaction to other HMG-CoA reductase inhibitors (statins).
* History of hypersensitivity reaction to inulin.
* Lipid-lowering drugs (including lipid lowering dietary supplements of food additives) within the last 4 weeks.
* Diabetes mellitus, defined as glycosylated hemoglobin (HbA1C) above the upper limit of normal (ULN).
* Uncontrolled arterial hypertension (>160/100mm Hg).
* Subjects considered to be unstable (event within 12 weeks) by the investigator after the following events: a myocardial infarction, unstable angina, myocardial revascularisation (PTCA, CABG surgery or another revascularisation procedure) or a transient ischaemic attack (TIA) or stroke.
* Significant arrythmias or conduction disturbances.
* Congestive heart failure (NYHA classes III or IV).
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception or have positive serum pregnancy test (a serum beta-human chorionic gonadotropin analysis).
* History of homozygous familial hypercholesterolaemia or known type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Use of concomitant medications.
* Current active liver disease(SGPT > 2xULN) or severe hepatic impairment.
* Unexplained serum CK > 3 times ULN (e.g. not due to recent trauma, intramuscular injections, heavy exercise etc.).
* Serum creatinine > 2,0 mg/dl and creatinine clearance <80ml/min.
* History of nephrolithiasis with calcium oxalate aggregation.
* Uncontrolled hypothyroidism defined as a thyroid stimulating hormone (TSH) > 1,5 times the UL or subjects whose thyroid replacement therapy was initiated within the last 3 month.
* Severe disorders of the gastrointestinal tract or other diseases which interfere with the pharmacodynamics and pharmacokinetics of the study drug.
* History of malignancy(unless a documented disease-free period exceeding 10 years is present) with the exception of basal cell or squamous cell carcinoma of the skin. Women with a history of cervical dysplasia would be permitted to enter the study provided they have 3 consecutive clear Papanicolaou (Pap) smears.
* History of organ allografts.
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subjects´s safety or successful participation in the trial.
* Participation in a clinical study within 4 weeks preceding treatment start.
* Past or present alcohol or drug abuse.
* Suspected or confirmed poor compliance.
* Previous enrolment in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Study Completion 2006-09

PRIMARY OUTCOMES:
Change in renal plasma flow from baseline in response to L-NMMA infusion after 6 weeks treatment with rosuvastatin.

SECONDARY OUTCOMES:
Change in renal plasma flow from baseline in response to L-NMMA infusion after 3 days treatment with rosuvastatin.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — CRC, Medizinsiche Klinik 4 - Nephrology and Hypertension, University of Erlangen-Nürnberg
Locations (1):
- CRC, Medizinische Klinik 4 - Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen, Krankenhausstrase 12, Germany

REFERENCES:
- [Result] Ott C, Schlaich MP, Schmidt BM, Titze SI, Schaufele T, Schmieder RE. Rosuvastatin improves basal nitric oxide activity of the renal vasculature in patients with hypercholesterolemia. Atherosclerosis. 2008 Feb;196(2):704-11. doi: 10.1016/j.atherosclerosis.2006.12.020. Epub 2007 Feb 12. PMID 17298834
- [Result] Ott C, Ritt M, Titze SI, Schaufele T, Schmieder RE. Rosuvastatin does not affect intrarenal hemodynamics in patients with hypercholesterolemia. J Nephrol. 2009 Sep-Oct;22(5):675-81. PMID 19810001
- [Result] Ott C, Schneider MP, Schlaich MP, Schmieder RE. Rosuvastatin improves pulse wave reflection by restoring endothelial function. Microvasc Res. 2012 Jul;84(1):60-4. doi: 10.1016/j.mvr.2012.03.007. Epub 2012 Mar 29. PMID 22484031
- [Result] Ott C, Raff U, Schneider MP, Titze SI, Schmieder RE. 25-hydroxyvitamin D insufficiency is associated with impaired renal endothelial function and both are improved with rosuvastatin treatment. Clin Res Cardiol. 2013 Apr;102(4):299-304. doi: 10.1007/s00392-012-0534-1. Epub 2012 Dec 21. PMID 23262496